CLINICAL TRIAL: NCT05079256
Title: A Preliminary Study on the Effect of Photothermal Laser Therapy on the Vascularization and Innervation of Psoriatic Lesions
Brief Title: Laser Induced Changes to Innervation and Vascularisation of Psoriatic Skin
Acronym: LPA-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nick van der Beek (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor-Investigator, Nick van der Beek, Managing director, ZBC MultiCare
Organization: ZBC MultiCare (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LPA-01
Record Dates: First submitted 2021-09-20; First posted 2021-10-15 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Lasers, Dye

STUDY DESIGN:
Intervention Model Description: single blinded intra-patient comparison
Masking Description: tissue samples are described using random pre-assigned codes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Laser therapy (Experimental): 595 nm Pulsed dye laser (PDL) therapy for psoriasis
  Interventions: Device: 595 nm Pulsed dye laser (Candela V-beam perfecta)

INTERVENTIONS:
Device: 595 nm Pulsed dye laser (Candela V-beam perfecta) — 595 nm pulsed dye laser therapy. 2 treatments Fluence ~ 6 - 9 J/cm^2 Pulse duration ~ 0.45 - 3.0 ms 33% overlap.

SUMMARY:
The researchers investigate the effect of a treatment with selective photothermolysis using a 595 nm pulsed dye laser on the blood vessel density and the nerve fibre density of a psoriatic lesion. By comparing tissue samples collected before and after two treatments, the researchers determine the relative effect of laser therapy on the (hyper)innervation of psoriatic skin.

DETAILED DESCRIPTION:
Vascular laser therapy for psoriasis seems to achieve a remarkably long treatment-free duration of remission. But why would sub-second heating of the blood vessels of the skin result in a year-long resolution of an infamously stubborn condition?

Unraveling the mechanism of action of laser therapy would not only allow for the improvement of existing laser therapy protocols but also, could open the door to a whole new range of interventions offering quasi-permanent solutions for patients. There is a high need for such enduring therapies: Psoriasis is both, a common and a costly skin condition. It affects between 1% and 9% of the population and has a very severe impact on the quality of life of the patient. It's chronic character implies lifelong treatment, and the associated risks and effort

This project aims to assess the effect of laser therapy on the blood vessels and (peripheral) innervation of psoriasis plaques. The primary objective is to quantify the regression and recovery of nerves compared to blood vessels. The researchers hypothesize that the recovery of nerves after Selective Photo Thermolysis (SPT) is decreased compared to the recovery of blood vessels.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 69 years of age
* Psoriasis vulgaris
* Skin type I - III
* Minimal surface of lesion of 3 cm2
* Contralateral psoriasis vulgaris lesions located on chest, back, or upper legs

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study if:

* The participant uses other treatments (than laser therapy) during the study or two weeks before the start of the study that are known to affect psoriasis
* The participant suffers from any known neurological, vascular, or immunological condition other than psoriasis.
* The participant is allergic to lidocaine

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2024-10-12 (Actual); Study Completion 2024-10-12 (Actual)

PRIMARY OUTCOMES:
Recovery ration | 6 months.
  Relative change in the ratio of the linear nerve density and linear blood vessel density.

SECONDARY OUTCOMES:
Recovery ratio vs lymphocyte infiltration | 6 months
  Correlation between change in the ratio of the linear nerve density and linear blood vessel density versus change in number of infiltrating lymphocytes
Clinical improvement | 6 months
  Change in severity determined using a visual-analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nick van der Beek, Ph.D, Principal Investigator — ZBC MultiCare
Locations (1):
- ZBC MultiCare, Hilversum, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
The data acquired during the investigation will be made available upon request.

REFERENCES:
- See also: This investigation is part of a larger research collaboration, more information on which can be found at the website mentioned above. — https://zbcmulticare.nl/lasering-psoriasis-away/